CLINICAL TRIAL: NCT00156468
Title: Office-Based Asthma Screening Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Halcyon Hill Foundation (Other); Robert Wood Johnson Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10035
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Behavioral: Provider Prompt

SUMMARY:
In prior work, we found that even children who have been seen by their physicians within the prior six months were frequently misclassified as having mild rather than persistent asthma. This study evaluations whether systematic office-based screening assists primary care physicians in identifying children with significant asthma and improves preventive care for asthma. We hypothesize that standardized screening in the office setting will improve the physician's ability to (a) identify children with significant asthma and (b) prescribe appropriate preventive medications.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 2-12
* Children arriving for an office visit in two Rochester, NY pediatric clinics
* Children with a prior diagnosis of asthma AND an exacerbation of symptoms within the previous 2 years

Exclusion Criteria:

* Children arriving at the office visit with an adult that is not their parent or guardian
* Children arriving at the office visit with a parent or guardian that does not speak English
* Children with other medical conditions making the assessment of asthma severity difficult (cystic fibrosis, heart conditions, etc.)

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 365
Dates: Start 2003-10; Study Completion 2005-09

PRIMARY OUTCOMES:
"Preventive Medication Actions (PMA)" taken by the provider at the time of the child's visit. A "PMA" is defined as a new medication prescription or change in medication dose.

SECONDARY OUTCOMES:
Alternate actions taken by the provider such as: discussion of environmental controls, medication refills, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jill S Halterman, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Background] Halterman JS, Kitzman H, McMullen A, Lynch K, Fagnano M, Conn KM, Yoos HL. Quantifying preventive asthma care delivered at office visits: the Preventive Asthma Care-Composite Index (PAC-CI). J Asthma. 2006 Sep;43(7):559-64. doi: 10.1080/02770900600859172. PMID 16939999
- [Background] Halterman JS, Fagnano M, Conn KM, Szilagyi PG. Do parents of urban children with persistent asthma ban smoking in their homes and cars? Ambul Pediatr. 2006 Mar-Apr;6(2):115-9. doi: 10.1016/j.ambp.2005.10.004. PMID 16530150
- [Result] Halterman JS, Fisher S, Conn KM, Fagnano M, Lynch K, Marky A, Szilagyi PG. Improved preventive care for asthma: a randomized trial of clinician prompting in pediatric offices. Arch Pediatr Adolesc Med. 2006 Oct;160(10):1018-25. doi: 10.1001/archpedi.160.10.1018. PMID 17018460